CLINICAL TRIAL: NCT02180204
Title: Phase IIb Study Comparing Tenecteplase to Alteplase in Acute Ischemic Stroke Within 3 to 4.5 Hours From Symptom Onset
Brief Title: Tenecteplase Versus Alteplase in Ischemic Stroke Management (TALISMAN)
Acronym: TALISMAN
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Reza Behrouz, DO (Other)
Responsible Party: Sponsor-Investigator, Reza Behrouz, DO, Associate Professor of Neurology, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013H000; TALISMAN (Other: The Ohio State University College of Medicine)
Record Dates: First submitted 2014-06-21; First posted 2014-07-02 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Ischemic Stroke
Keywords: Cerebral Infarction; Ischemic Stroke; Thrombolysis
MeSH Terms: conditions — Ischemic Stroke; Cerebral Infarction | interventions — Tenecteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tenecteplase (Experimental): Tenecteplase 0.25 mg/kg IV - Maximum dose: 25 mg
  Interventions: Drug: Tenecteplase
- Alteplase (Active Comparator): Alteplase 0.9 mg/kg IV - Maximum dose: 90 mg
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Tenecteplase — Tenecteplase 0.25 mg/kg IV - Maximum 25 mg
  Other Names: TNKase
  Arms: Tenecteplase
Drug: Alteplase — Alteplase 0.9 mg/kg IV - Maximum: 90 mg
  Other Names: Activase; t-PA
  Arms: Alteplase

SUMMARY:
This is a double-blind parallel arm randomized trial aimed to assess efficacy and safety of intravenous Tenecteplase compared to intravenous Alteplase in eligible patients who present with symptoms of acute ischemic stroke within 3 to 4.5 hours from onset.

DETAILED DESCRIPTION:
Patients presenting with symptoms of acute ischemic stroke (AIS) who present within 3 to 4.5 hours of symptom onset and who meet the inclusion criteria for intravenous (IV) thrombolysis will receive, in a randomized, double-blind fashion, either IV Alteplase at 0.9 mg/kg per standard protocol or IV Tenecteplase at 0.25 mg/kg with saline infusion over one hour. Patients must also have no exclusion criteria for IV thrombolysis within the 3 to 4.5 hour window. The only required imaging is non-contrasted CT of the head. Patients will be monitored according to standard post-thrombolytic care. A CT of the head will be performed at 24 hours based on standard protocol or if there is any neurological change. Neurological function at 24 hours using NIHSS and at 3 months based on modified mRS and the NIHSS.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years
2. Acute neurologic deficit with an NIHSS ≥ 4
3. Non-enhanced computed tomography (NECT) of the head showing no hemorrhage
4. Acute ischemic stroke symptoms with onset, or time last known well, clearly defined between 3 and 4.5 hours
5. Treatment can be initiated within 3 to 4.5 hours from symptom onset

Exclusion Criteria:

1. Evidence of intracranial hemorrhage on NECT
2. Clinical suspicion of subarachnoid hemorrhage even with normal NECT
3. NECT shows hypo-density greater than 1/3 cerebral hemisphere)
4. History of intracranial hemorrhage/stroke
5. Uncontrolled HTN: At time treatment begins SBP remains >185 mmHg or DBP remains >110 mmHg despite repeated measurements
6. Known arteriovenous malformation, neoplasm, or aneurysm
7. Witnessed seizure at stroke onset
8. Acute bleeding tendencies
9. Platelet count <100,000/mm3
10. Heparin received in prior 48 hours with elevated aPTT
11. Current use of an anticoagulant (Coumadin/Warfarin) irrespective of INR
12. Prior use (within 48 hours) of direct thrombin inhibitors (dabigatran) or direct factor Xa inhibitors (rivaroxaban, apixaban)
13. Within prior 3 months: intracranial or spinal surgery, head trauma, or previous stroke
14. Arterial puncture at non-compressible site within last 7 days
15. Woman of child bearing age who has a positive pregnancy test
16. NIH stroke scale >25 (severe deficit) or <4 and no dysphasia (mild deficit) or rapidly improving
17. Symptoms spontaneously clearing
18. 14 days post-operative or post major trauma
19. Recent gastrointestinal or urinary tract hemorrhage within the past 21 days
20. Recent acute MI within the past 3 months
21. Serum glucose <50 mg/dl or >400 mg/dL
22. Age >80 or less than 18
23. History of ischemic stroke AND diabetes mellitus
24. Unable to obtain consent from patient or power of attorney
25. Baseline mRS > 2
26. Consent not obtained by 20 minutes prior to closure of the therapeutic window.
27. The subject has been treated with a thrombolytic agent within the past 72 hours
28. The subject is a pregnant woman (positive serum βHCG pregnancy test, positive urine pregnancy test or clinically evident pregnancy)
29. The subject is, in the opinion of the investigator, unlikely to comply with the clinical study protocol or is unsuitable for any other reason

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Neurological outcome | 90 days
  Measured by modified Rankin Scale score

SECONDARY OUTCOMES:
Symptomatic intracranial hemorrhage | 24 hours
  Twenty-four hour brain CT scan showing intracranial hemorrhage in conjuction with neurological deterioration of 4 points or more on the NIHSS

CONTACTS AND LOCATIONS:
Overall Officials: Reza Behrouz, DO, Principal Investigator — The Ohio State University College of Medicine
Locations (1):
- The Ohio State University College of Medicine, Columbus, Ohio, United States

REFERENCES:
- [Background] Parsons M, Spratt N, Bivard A, Campbell B, Chung K, Miteff F, O'Brien B, Bladin C, McElduff P, Allen C, Bateman G, Donnan G, Davis S, Levi C. A randomized trial of tenecteplase versus alteplase for acute ischemic stroke. N Engl J Med. 2012 Mar 22;366(12):1099-107. doi: 10.1056/NEJMoa1109842. PMID 22435369
- [Background] Parsons MW, Miteff F, Bateman GA, Spratt N, Loiselle A, Attia J, Levi CR. Acute ischemic stroke: imaging-guided tenecteplase treatment in an extended time window. Neurology. 2009 Mar 10;72(10):915-21. doi: 10.1212/01.wnl.0000344168.05315.9d. PMID 19273826
- [Background] Haley EC Jr, Thompson JL, Grotta JC, Lyden PD, Hemmen TG, Brown DL, Fanale C, Libman R, Kwiatkowski TG, Llinas RH, Levine SR, Johnston KC, Buchsbaum R, Levy G, Levin B; Tenecteplase in Stroke Investigators. Phase IIB/III trial of tenecteplase in acute ischemic stroke: results of a prematurely terminated randomized clinical trial. Stroke. 2010 Apr;41(4):707-11. doi: 10.1161/STROKEAHA.109.572040. Epub 2010 Feb 25. PMID 20185783
- [Background] Haley EC Jr, Lyden PD, Johnston KC, Hemmen TM; TNK in Stroke Investigators. A pilot dose-escalation safety study of tenecteplase in acute ischemic stroke. Stroke. 2005 Mar;36(3):607-12. doi: 10.1161/01.STR.0000154872.73240.e9. Epub 2005 Feb 3. PMID 15692126
- [Background] Lees KR, Bluhmki E, von Kummer R, Brott TG, Toni D, Grotta JC, Albers GW, Kaste M, Marler JR, Hamilton SA, Tilley BC, Davis SM, Donnan GA, Hacke W; ECASS, ATLANTIS, NINDS and EPITHET rt-PA Study Group; Allen K, Mau J, Meier D, del Zoppo G, De Silva DA, Butcher KS, Parsons MW, Barber PA, Levi C, Bladin C, Byrnes G. Time to treatment with intravenous alteplase and outcome in stroke: an updated pooled analysis of ECASS, ATLANTIS, NINDS, and EPITHET trials. Lancet. 2010 May 15;375(9727):1695-703. doi: 10.1016/S0140-6736(10)60491-6. PMID 20472172
- [Background] Behrouz R. Intravenous tenecteplase in acute ischemic stroke: an updated review. J Neurol. 2014 Jun;261(6):1069-72. doi: 10.1007/s00415-013-7102-0. Epub 2013 Sep 15. PMID 24036924
- [Derived] Logallo N, Kvistad CE, Thomassen L. Therapeutic Potential of Tenecteplase in the Management of Acute Ischemic Stroke. CNS Drugs. 2015;29(10):811-8. doi: 10.1007/s40263-015-0280-9. PMID 26387127